CLINICAL TRIAL: NCT00794222
Title: A Randomised Controlled Trial Investigating a Mobile Phone Self-monitoring Tool (Mobiletype) to Increase Emotional Self-awareness and Reduce Depressive Symptoms in Young People.
Brief Title: A Mobile Phone Self-Monitoring Tool to Increase Emotional Self-Awareness and Reduce Depression in Young People
Acronym: mobiletype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RCH28113
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Depression
Keywords: Cellular phones; mental health; Early intervention; prevention; momentary sampling; Adolescent
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mood monitoring (Experimental): The mobiletype monitoring intervention group will monitor their current activities, current mood, responses to negative mood, any recent stressors and coping strategies. Other activities monitored include eating patterns, exercise patterns, quantity and quality of sleep and alcohol and cannabis use.
  Interventions: Device: Mobile Tracking Young People's Experiences (mobiletype)
- Comparison monitoring program (No Intervention): The mobiletype monitoring comparison group will monitor their current activities, eating patterns, exercise patterns, quantity and quality of sleep and alcohol and cannabis use.
  This program excludes questions about mood, stress and coping strategies.

INTERVENTIONS:
Device: Mobile Tracking Young People's Experiences (mobiletype) — A mobile phone self-monitoring program, based on momentary sampling techniques, that prompts young people to complete it four times a day. The program asks several questions about daily activities, mood, stress, eating and exercise.
  Arms: Mood monitoring

SUMMARY:
The mobiletype program is a mental health assessment and monitoring tool that runs on mobile phones.

The program assesses the general mental health of young people in real-time and transmits this data to a website to be reviewed by their general practitioner (GP) in consultation with their patient. The website consists of individualised feedback reports for each participant, and graphical displays of the monitoring data. The primary aims of the current project are to examine: (1) whether the process of self-monitoring via the mobiletype program increases young people's awareness of their mood and reduces depressive symptoms and (2) whether emotional self-awareness mediates the relationship between self-monitoring and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 - 24 years of age
* Proficient English
* Patients must be deemed to have an emotional/mental health concern by their GP or be screened to have at least a mild mental health problem (a score of 16 or above) on the K10 Symptom Scale

Exclusion Criteria:

* Severe psychiatric or medical condition that prevents the person from complying with either the requirements of informed consent or the study protocol.
* Young people referred to a mental health specialist by their GP will be excluded only if they obtain a specialist appointment during the mobiletype study period (2 - 4 weeks).

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Pre-, post-monitoring, 6-week follow up & 6 month follow-up
Emotional Self Awareness | Pre-, post-, 6-weeks post- and 6-months post-test

SECONDARY OUTCOMES:
Detection of mental health problems | Pre-, post-monitoring, 6 week and 6 month follow up
Pathways to care | Pre-, post-monitoring, 6 week and 6 month follow up
Patient's satisfaction with their GP | Pre-, post-monitoring, 6 week and 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia D Kauer, BBSci(Hons), Principal Investigator — Murdoch Childrens Research Instititue; Sophie C Reid, PhD,MPsych, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Clifton Hill Medical Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Reid SC, Kauer SD, Hearps SJ, Crooke AH, Khor AS, Sanci LA, Patton GC. A mobile phone application for the assessment and management of youth mental health problems in primary care: health service outcomes from a randomised controlled trial of mobiletype. BMC Fam Pract. 2013 Jun 19;14:84. doi: 10.1186/1471-2296-14-84. PMID 23782796
- [Derived] Kauer SD, Reid SC, Crooke AH, Khor A, Hearps SJ, Jorm AF, Sanci L, Patton G. Self-monitoring using mobile phones in the early stages of adolescent depression: randomized controlled trial. J Med Internet Res. 2012 Jun 25;14(3):e67. doi: 10.2196/jmir.1858. PMID 22732135
- [Derived] Reid SC, Kauer SD, Hearps SJ, Crooke AH, Khor AS, Sanci LA, Patton GC. A mobile phone application for the assessment and management of youth mental health problems in primary care: a randomised controlled trial. BMC Fam Pract. 2011 Nov 29;12:131. doi: 10.1186/1471-2296-12-131. PMID 22123031